CLINICAL TRIAL: NCT03061721
Title: A Phase 2, Prospective, Multicenter, Double-blind, Randomized Study of Saroglitazar Magnesium 1 mg, 2 mg or 4 mg Versus Placebo in Patients With Nonalcoholic Fatty Liver Disease and/or Nonalcoholic Steatohepatitis
Brief Title: Saroglitazar Magnesium in Patients With Nonalcoholic Fatty Liver Disease and/or Nonalcoholic Steatohepatitis
Acronym: EVIDENCES IV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SARO.16.005
Record Dates: First submitted 2017-02-07; First posted 2017-02-23 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
Keywords: NASH; NAFLD; Saroglitazar
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — saroglitazar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Saroglitazar magnesium 1 mg (Experimental): Saroglitazar magnesium 1 mg tablet orally once daily in the morning before breakfast for 16 weeks.
  Interventions: Drug: Saroglitazar magnesium 1 mg
- Saroglitazar magnesium 2 mg (Experimental): Saroglitazar magnesium 2 mg tablet orally once daily in the morning before breakfast for 16 weeks.
  Interventions: Drug: Saroglitazar magnesium 2 mg
- Saroglitazar magnesium 4 mg (Experimental): Saroglitazar magnesium 4 mg tablet orally once daily in the morning before breakfast for 16 weeks.
  Interventions: Drug: Saroglitazar magnesium 4 mg
- Placebos (Placebo Comparator): Placebo tablet orally once daily in the morning before breakfast for 16 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Saroglitazar magnesium 1 mg — Patients randomly assigned to this group will receive Saroglitazar magnesium 1 mg tablet orally once daily for 16 weeks.
  Arms: Saroglitazar magnesium 1 mg
Drug: Saroglitazar magnesium 2 mg — Patients randomly assigned to this group will receive Saroglitazar magnesium 2 mg tablet orally once daily for 16 weeks.
  Arms: Saroglitazar magnesium 2 mg
Drug: Saroglitazar magnesium 4 mg — Patients randomly assigned to this group will receive Saroglitazar magnesium 4 mg tablet orally once daily for 16 weeks.
  Arms: Saroglitazar magnesium 4 mg
Drug: Placebos — Patients randomly assigned to this group will receive placebo tablet orally once daily for 16 weeks.
  Arms: Placebos

SUMMARY:
This is a randomized, double-blind, placebo-controlled study in up to 104 patients with a diagnosis of Non-alcoholic fatty Liver disease (NAFLD) and/or Non-alcoholic steatohepatitis (NASH). The study will be conducted over a period of up to 22 weeks and will include an optional Prescreening, Screening (Days -35 to -7) Phase, a 16-week Treatment Phase following randomization on Day 1. Patients will be randomly assigned in a ratio of 1:1:1:1 to receive Saroglitazar Magnesium 1mg or 2 mg or 4 mg or matching placebo once daily in the morning before breakfast for 16 Weeks. The primary endpoint of the study is percentage change from baseline in serum Alanine transaminase (ALT) levels at Week 16 in the Saroglitazar Magnesium groups as compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18 to 75 years of age, with body mass index (BMI) ≥ 25 kg/m^2.
2. Documented diagnosis of NAFLD established either by imaging (ultrasound, computed tomography [CT] scan or Magnetic resonance imaging [MRI]) or liver biopsy showing NASH or simple steatosis, within the 24 months preceding Visit 1. The diagnosis of NAFLD is made according to the American Association for the Study of Liver Diseases (AASLD) criteria (Chalasani et al. Hepatology 2012; 55:2005-2023).
3. ALT level of ≥50 U/L at Visit 1 and Visit 2 with ≤30% variance between the levels at Visit 1 and Visit 2.
4. Patient's demonstration of understanding of study requirements and treatment procedures, willingness to comply with all protocol-required evaluations; provision of written informed consent before any study specific tests or procedures are performed.

Exclusion Criteria:

1. Consumption of > 3 units of alcohol per day (> 21 units per week) if male and > 2 units of alcohol per day (>14 units per week) if female for at least 3 consecutive months in the 5 years preceding Visit 1 (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor).
2. Presence of alternative causes of fatty liver, including:

   1. Weight change >5% within the 3 months preceding Visit 1
   2. Total parenteral nutrition, starvation or protein-calorie malnutrition within the 90 days preceding Visit 1.
   3. Use of drugs associated with NAFLD for more than 12 consecutive weeks in the 1 year before Visit 1, including amiodarone, tamoxifen, methotrexate, systemic glucocorticoids, anabolic steroids, tetracycline, estrogens in doses higher than used in oral contraceptives, vitamin A, L asparaginase, valproate, chloroquine or antiretroviral drugs
3. Initiation of vitamin E at doses > 100 IU/day, or multivitamins containing > 100 IU/day of vitamin E in the 3 months preceding Visit 1.
4. Use of drugs with potential effect on NASH such as ursodeoxycholic acid, S-adenosylmethionine (SAM-e), betaine, pentoxifylline, obeticholic acid or milk thistle in the 3 months prior to Visit 1.
5. Changing doses of statins (simvastatin, pitavastatin, pravastatin, atorvastatin, fluvastatin, lovastatin, rosuvastatin) or fibrates (clofibrate, fenofibrate) in the 3 months preceding Visit 1.
6. Use of thiazolidinediones (pioglitazone, rosiglitazone).
7. Use of drugs that are known Cytochrome P4502C8 (CYP2C8) inhibitors/substrate
8. History of bowel surgery (gastrointestinal (bariatric) surgery or undergoing evaluation for bariatric surgery for obesity, extensive small-bowel resection or orthotopic liver transplant (OLT) or listed for OLT.
9. History of other chronic liver disease (chronic hepatitis C, (HCV) infection, irrespective of their mRNA HCV assay status or active hepatitis B infection, (i.e., serum positive for hepatitis B surface antigen) or autoimmune hepatitis, cholestatic and metabolic liver diseases) or hemochromatosis
10. Patient has known cirrhosis, either based on clinical criteria or liver histology.
11. Patient with Internation Normalised Ratio (INR) >1.3.
12. Type 1 diabetes mellitus.
13. Poorly controlled type 2 diabetes mellitus, i.e., glycosylated hemoglobin (HbA1c) > 9%.
14. Unstable cardiovascular disease, including:

    1. unstable angina, (i.e., new or worsening symptoms of coronary heart disease within the 3 months preceding Visit 1), acute coronary syndrome within the 6 months preceding Visit 1, acute myocardial infarction within the 3 months preceding Visit 1 or heart failure of New York Heart Association class (III - IV) or worsening congestive heart failure, or coronary artery intervention, within the 6 months preceding Visit 1
    2. history of (within 3 months preceding Visit 1) or current unstable cardiac dysrhythmias
    3. uncontrolled hypertension (systolic blood pressure [BP] > 160 mmHg and/or diastolic BP > 100 mmHg)
    4. stroke or transient ischemic attack within the 6 months preceding Visit 1.
15. History of myopathies or evidence of active muscle disease.
16. History of malignancy in the 5 years preceding Visit 1 and/or active neoplasm with the exception of resolved superficial nonmelanoma skin cancer.
17. Any of the following laboratory values:

    1. Hemoglobin < 9 g/dL
    2. White blood cell count < 2.5 × 103/μL
    3. Neutrophil count < 1.5 × 103/μL
    4. Platelets < 100 × 103/μL
    5. Total Serum bilirubin > 1.5 mg/dL (except in patient with known Gilbert bilirubin where Total Bilirubin up to 2.5 mg/dL is allowed), if it is <1.5 mg/dL at screening and >30% variance in the levels at Visit 1 and Visit 2
    6. Albumin < 3.2 g/dL
    7. Serum creatinine >1.5 mg/dL
    8. Serum ALT or Aspartate aminotransferase (AST) > 250 IU/L at Visit 1 or Visit 2 .
18. Contraindications to Saroglitazar Magnesium or has any conditions affecting the ability to evaluate the effects of Saroglitazar Magnesium.
19. Known allergy, sensitivity or intolerance to the study drug, placebo or formulation ingredients.
20. Participation in any other therapeutic clinical study within the 3 months preceding Visit 1, including participation in any other NAFLD/NASH clinical trials.
21. History of bladder disease and/or hematuria or has current hematuria except due to a urinary tract infection.
22. Illicit substance abuse within the 12 months preceding Visit 1.
23. Pregnancy-related exclusions, including:

    1. Pregnant/lactating female (including a positive serum pregnancy test at Visit 1)
    2. A male patient has to use a condom with spermicide, and the female partner of the male patient has to use an intrauterine device OR a diaphragm with spermicide OR oral contraceptive pills.
    3. If a male patient has undergone a vasectomy, the female partner does not have to use any contraception.
    4. A female patient has to use either an intrauterine device OR a diaphragm with spermicide OR oral contraceptive pills. The male partner of the female patient has to use a condom with spermicide.
    5. If the female patient is surgically sterilized for at least the 6 months preceding Visit 1 or postmenopausal, defined as at least 12 months with no menses and without an alternative cause, the male partner of the female patient does not have to use any contraception.
24. History or other evidence of severe illness or any other conditions that would make the patient, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease, HIV, coronary artery disease or active gastrointestinal conditions that might interfere with drug absorption).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deven V Parmar, MD,FACP,FCP, Study Director — Zydus Therapeutics Inc.
Locations (18):
- United States (18):
  - Precision Research, Chula Vista, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - California liver research institute, Pasadena, California
  - Precision Research, San Diego, California
  - University of Florida, Gainesville, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Avail Clinical Research, Orange City, Florida
  - Indiana University, Indianapolis, Indiana
  - Mercy Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Awasty Research Network, LLC, Marion, Ohio
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - AIG Research, Hermitage, Tennessee
  - Liver Consultants, Dallas, Texas
  - The Liver Institute, San Antonio, Texas
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Result] Gawrieh S, Noureddin M, Loo N, Mohseni R, Awasty V, Cusi K, Kowdley KV, Lai M, Schiff E, Parmar D, Patel P, Chalasani N. Saroglitazar, a PPAR-alpha/gamma Agonist, for Treatment of NAFLD: A Randomized Controlled Double-Blind Phase 2 Trial. Hepatology. 2021 Oct;74(4):1809-1824. doi: 10.1002/hep.31843. Epub 2021 Jul 19. PMID 33811367
- [Derived] Siddiqui MS, Parmar D, Sheikh F, Sarin SK, Cisneros L, Gawrieh S, Momin T, Duseja A, Sanyal AJ. Saroglitazar, a Dual PPAR alpha/gamma Agonist, Improves Atherogenic Dyslipidemia in Patients With Non-Cirrhotic Nonalcoholic Fatty Liver Disease: A Pooled Analysis. Clin Gastroenterol Hepatol. 2023 Sep;21(10):2597-2605.e2. doi: 10.1016/j.cgh.2023.01.018. Epub 2023 Jan 31. PMID 36731585
- See also: Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of — http://pubmed.ncbi.nlm.nih.gov/22488764/
- See also: Gawrieh S, Noureddin M, Loo N, Mohseni R, Awasty V, Cusi K, Kowdley KV, Lai M, Schiff E, Parmar D, Patel P, Chalasani N. Saroglitazar, a PPAR-alpha/gamma Agonist, for Treatment of NAFLD: A Randomized Controlled Double-Blind Phase 2 Trial. — http://pubmed.ncbi.nlm.nih.gov/33811367/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebos
Started | 26 | 25 | 27 | 28
Completed | 26 | 20 | 27 | 25
Not Completed | 0 | 5 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebos | Total
Number analyzed (Participants) | 26 | 25 | 27 | 28 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (12.89) | 47.9 (10.44) | 49 (10.97) | 48.7 (10.46) | 49.2 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 12 | 13 | 50
  Male | 13 | 13 | 15 | 15 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 12 | 13 | 43
  Not Hispanic or Latino | 16 | 17 | 15 | 15 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 3 | 3 | 3 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 22 | 21 | 24 | 24 | 91
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.630 (4.2451) | 35.702 (8.5653) | 32.489 (5.1611) | 33.809 (4.4599) | 33.875 (5.8374)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Serum Alanine Aminotransferase (ALT) Levels at Week 16
Description: Percentage change from baseline in serum ALT levels at Week 16 in the Saroglitazar Magnesium groups as compared to the placebo group
Time Frame: Baseline and Week 16
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- Placebo: Placebo tablet orally once daily in the morning before breakfast for 16 weeks.
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 26 | 25 | 27 | 28
Percentage change | -26.2 (33.36) | -27.0 (26.52) | -44.9 (26.26) | 2.6 (32.06)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 1 mg vs Placebo; Test type: Superiority; p = 0.0002, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Superiority; p = 0.0001, ANCOVA
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

2. Secondary Outcome: Change in Liver Fat Content as Measured by Magnetic Resonance Imaging-derived Proton Density-fat Fraction (MRI-PDFF)
Description: Change in liver fat content as measured by magnetic resonance imaging-derived proton in Saroglitazar Magnesium groups as compared to the placebo group
Time Frame: Baseline and Week 16
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of Liver fat
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 26 | 25 | 27 | 28
percentage of Liver fat | 0.53 (5.228) | -0.36 (4.297) | -4.21 (6.231) | -0.28 (5.409)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 1 mg vs Placebo; Test type: Superiority; p = 0.5681, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Superiority; p = 0.4487, ANCOVA
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.0021, ANCOVA

3. Secondary Outcome: Proportion of Patients With Sustain Decrease in Serum ALT Levels
Description: Proportion of patients with sustain decrease in serum ALT levels in Saroglitazar Magnesium groups as compared to the placebo group
Time Frame: Week 16
Population: Full Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 26 | 25 | 27 | 28
Participants | 22 | 22 | 26 | 14
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 1 mg vs Placebo; Test type: Superiority; p = 0.0070, Chi-squared
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Superiority; p = 0.0031, Chi-squared
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.0001, Chi-squared

4. Secondary Outcome: Changes in Cytokeratin-18
Description: Changes in cytokeratin-18 in Saroglitazar Magnesium groups as compared to the placebo group
Time Frame: baseline and Week 16
Population: full analysis set
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 25 | 23 | 27 | 25
U/L | -3.0 (693.75) | -330.3 (590.37) | -64.1 (303.59) | 97.4 (437.10)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 1 mg vs Placebo; Test type: Superiority; p = 0.2241, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Superiority; p = 0.0304, ANCOVA
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.0595, ANCOVA

5. Secondary Outcome: Changes in Enhanced Liver Fibrosis
Description: Changes in enhanced liver fibrosis in Saroglitazar Magnesium groups as compared to the placebo group The ELF Score is a liver fibrosis score that is calculated by use of an algorithm: ELF score score = -7.412 + (ln(HA)*0.681) + (ln(P3NP)*0.775) + (ln(TIMP1)*0.494).
  HA=hyaluronic acid concentration P3NP=procollagen 3 amino terminal peptide concentration TIMP1=tissue inhibitor matrix metalloproteinase 1 concentration. All are measured in serum.
  The ELF score has been reported to show good correlations with fibrosis stages in chronic liver disease, with higher ELF scores associated with higher fibrosis stages. The ELF score is hence used as a prognostic marker for disease progression: ELF score < 9.8 : Low risk of progression, ELF score 9.8 to < 11.3 : Moderate risk of progression and ELF score > = 11.3 : High risk of progression
Time Frame: baseline and Week 16
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 26 | 25 | 27 | 28
units on a scale | -0.2 (0.78) | -0.3 (0.86) | -0.3 (0.72) | 0.4 (0.78)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 1 mg vs Placebo; Test type: Superiority; p = 0.0449, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Superiority; p = 0.0053, ANCOVA
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.0036, ANCOVA

6. Secondary Outcome: Change in Aspartate Aminotransferase-to-platelet Ratio Index
Description: Change in aspartate aminotransferase-to-platelet ratio index in Saroglitazar Magnesium groups as compared to the placebo group APRI was calculated as ([AST level/AST upper limit of normal]/ [Platelet count 1^09/L]) ×100, where AST is aspartate aminotransferase. The aspartate transaminase to platelet ratio index (APRI) is used to assess the risk of liver fibrosis.
  Higher APRI score represents a higher risk of liver fibrosis
Time Frame: Baseline and Week 16
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 26 | 25 | 27 | 28
units on a scale | -0.3 (0.56) | -0.2 (0.51) | -0.3 (0.47) | 0.1 (0.73)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 1 mg vs Placebo; Test type: Superiority; p = 0.0045, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Superiority; p = 0.0026, ANCOVA
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.0004, ANCOVA

7. Secondary Outcome: Pharmacokinetics of Saroglitazar Magnesium: Maximum Plasma Concentration (Cmax)
Description: Maximum plasma concentration (Cmax) of Saroglitazar
Time Frame: PK sampling timepoints: Pre-dose (0.0), 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, and 24 hours post-dose of Visit 7 (Week 16)
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 5 | 6 | 8
ng/mL | 65.034 (17.579) | 98.995 (77.189) | 219.475 (111.521)

8. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Time to reach maximum plasma concentration (Tmax) of saroglitazar
Time Frame: as for outcome 7
Population: PK population
Measure: Median (Full Range); unit: hours
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 5 | 6 | 8
hours | 0.920 [0.500 to 1.020] | 1.500 [1.000 to 3.000] | 0.990 [0.500 to 2.080]

9. Secondary Outcome: Terminal Half-life (t1/2)
Description: Terminal Half-life (t1/2) of saroglitazar
Time Frame: as for outcome 7
Population: PK population For Saroglitazar 4 mg, one subject was not considered for calculation of Half-life as adjusted R square was observed <0.8000 and AUC_%Extrap_obs>20%. Hence, N=07 instead of 08 for Half-life
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 5 | 6 | 7
hour | 6.040 (1.314) | 6.597 (4.217) | 5.429 (1.509)

10. Secondary Outcome: Area Under the Curve From the Time of Dosing to the Last Measurable Concentration (AUC0-t)
Description: Area under the curve from the time of dosing to the last measurable concentration for saroglitazar
Time Frame: PK sampling timepoints: Pre-dose (0.0), 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, and 24 hours post-dose of Visit 3 (Week 0)
Population: PK population
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 5 | 6 | 8
hr*ng/mL | 171.064 (45.818) | 301.227 (202.061) | 667.646 (175.024)

11. Secondary Outcome: Area Under the Curve From the Time of Dosing to the Infinity (AUC 0-inf)
Description: Area under the curve from the time of dosing to the infinity (AUC 0-inf) for Saroglitazar
Time Frame: as for outcome 10
Population: PK population For Saroglitazar 4 mg, one subject was not considered for calculation of AUC 0-inf as adjusted R square was observed <0.8000 and AUC_%Extrap_obs>20%. Hence, N=07 instead of 08 for AUC 0-inf
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 4 | 6 | 7
hr*ng/mL | 167.735 (45.322) | 305.532 (203.074) | 652.497 (169.565)

12. Secondary Outcome: Elimination Rate Constant (λz)
Description: Elimination rate constant (λz) for saroglitazar
Time Frame: as for outcome 7
Population: PK population For Saroglitazar 4 mg, one subject was not considered for calculation of Kel as adjusted R square was observed <0.8000 and AUC_%Extrap_obs>20%. Hence, N=07 instead of 08 for Kel
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 5 | 6 | 7
per hour | 0.119 (0.027) | 0.129 (0.047) | 0.136 (0.035)

13. Secondary Outcome: Apparent Volume of Distribution (Vd/F)
Description: Apparent volume of distribution (Vd/F) for Saroglitazar
Time Frame: as for outcome 7
Population: PK population For Saroglitazar 4 mg, one subject was not considered for calculation of Vd/F as adjusted R square was observed <0.8000 and AUC_%Extrap_obs>20%. Hence, N=07 instead of 08 for Vd/F
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 5 | 6 | 7
mL | 49788.200 (18040.188) | 81341.167 (72030.406) | 53772.143 (17575.770)

14. Secondary Outcome: Apparent Clearance (CL/F)
Description: Apparent clearance (CL/F) for Saroglitazar
Time Frame: as for outcome 7
Population: PK population For Saroglitazar 4 mg, one subject was not considered for calculation of CL/F as adjusted R square was observed <0.8000 and AUC_%Extrap_obs>20%. Hence, N=07 instead of 08 for CL/F.
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 5 | 6 | 7
mL/hour | 5969.472 (2502.313) | 8030.060 (2356.620) | 6972.059 (1890.090)

15. Secondary Outcome: Change in Quality of Life Assessed by the Short-Form 36 Health Survey
Description: Quality of life will be assessed by the Short-Form 36 Health Survey The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (domains) as well as psychometrically based physical and mental health summary measures. The SF-36 taps 8 health concepts: physical functioning, bodily pain, physical role functioning, emotional role functioning, emotional well-being, social functioning, vitality, and general health perceptions. The 8 scales are further summarized to 2 distinct higher-ordered clusters: the PCS and mental composite t-score (MCS). The range for all 8 domains as well as for the composite t-scores is from 0 to 100 with 100 as best possible health status and 0 as worst health status.
Time Frame: baseline and 16 Week
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 26 | 25 | 27 | 28
units on a scale | -1.7 (7.24) | -2.2 (7.57) | -3.8 (10.77) | -1.0 (6.16)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 1 mg vs Placebo; Test type: Superiority; p = 0.2387, ANCOVA
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Superiority; p = 0.1496, ANCOVA
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.0445, ANCOVA

16. Secondary Outcome: Safety and Tolerability of Saroglitazar Magnesium
Description: Number of participants with adverse events
Time Frame: Baseline to Week 17
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebos
Number analyzed (Participants) | 26 | 25 | 27 | 28
participants | 13 | 13 | 14 | 19

ADVERSE EVENTS:
Time Frame: 16 Weeks
Arm/Group | Saroglitazar Magnesium 1 mg | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebos
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/25 | 1/27 | 0/28
Other Adverse Events (participants affected / at risk) | 7/26 | 6/25 | 3/27 | 5/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saroglitazar Magnesium 1 mg (N=26) | Saroglitazar Magnesium 2 mg (N=25) | Saroglitazar Magnesium 4 mg (N=27) | Placebos (N=28)
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Mental Status Change (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saroglitazar Magnesium 1 mg (N=26) | Saroglitazar Magnesium 2 mg (N=25) | Saroglitazar Magnesium 4 mg (N=27) | Placebos (N=28)
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 3 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT03061721/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT03061721/SAP_001.pdf